CLINICAL TRIAL: NCT02128074
Title: A Phase 2 Pilot Study of KRX-0502 (Ferric Citrate) in Treating Iron-deficiency Anemia in Patients With Stage 3-5 Non-dialysis Dependent Chronic Kidney Disease (NDD-CKD)
Brief Title: A Pilot Study of KRX-0502 (Ferric Citrate, Administered Without Food, in Treating Iron-deficiency Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRX-0502-207
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-11

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KRX-0502 (Experimental): KRX-0502 (ferric citrate)
  Interventions: Drug: KRX-0502

INTERVENTIONS:
Drug: KRX-0502 — 1g tablets of KRX-0502
  Other Names: ferric citrate

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of KRX-0502, administered without food, in treating iron deficiency anemia in subjects with stage 3 to 5 non-dialysis dependent chronic kidney disease (NDD-CKD).

DETAILED DESCRIPTION:
Previous clinical trials have tested KRX-0502 administered with food, in dialysis-dependent and NDD-CKD patients.

This clinical trial will evaluate the safety and efficacy of KRX-0502 in treating iron deficiency anemia in anemic, stage III to V NDD-CKD patients in a new dosing regimen (without food).

ELIGIBILITY:
Inclusion Criteria:

* Males and non-lactating females with negative serum pregnancy test (for females of child-bearing potential) at Screening
* Age ≥ 18 years
* Serum ferritin ≤ 300 ng/mL and TSAT ≤ 25% at Screening
* Hemoglobin ≥9.0 g/dL and ≤11.5 g/dL at Screening
* eGFR <60 mL/min at Screening using the 4-variable Modification of Diet in Renal Disease (MDRD) equation

Exclusion Criteria:

* Subjects receiving phosphate binder medication(s) at, or within 4 weeks prior to, screening
* Symptomatic gastrointestinal bleeding, inflammatory bowel disease, inflammatory bowel syndrome and/or Crohn's Disease within 24 weeks prior to \ Screening
* Evidence of acute kidney injury or requirement for dialysis within 8 weeks prior to Screening
* Kidney transplant anticipated or start of dialysis expected within 16 weeks of Screening
* History of hemochromatosis
* IV iron administered within 4 weeks prior to Screening
* Erythropoiesis-Stimulating Agent (ESA) administered within 4 weeks prior to Screening
* Blood transfusion within 4 weeks prior to Screening
* Receipt of any investigational drug within 4 weeks prior to Screening
* Cause of anemia other than iron deficiency or chronic kidney disease
* History of malignancy in the last five years
* Active drug or alcohol dependence or abuse (excluding tobacco use) within the 12 months prior to Screening
* Any known allergies to iron products
* Previous intolerance to oral ferric citrate
* Psychiatric disorder that interferes with the subject's ability to comply with the study protocol
* Planned surgery or hospitalization during the trial
* Any other medical condition that, in the opinion of the PI, renders the subject unable to or unlikely to complete the trial or that would interfere with optimal participation in the trial or produce significant risk to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Yagil, MD, Study Chair — The Barzilai Medical Center
Locations (3):
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Western Galilee Hospital, Nahariya
  - Nazareth Hospital- EMMS, Nazareth

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KRX-0502
Started | 32
Completed | 26
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | KRX-0502
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin From Baseline to the End of 8-week Treatment Period
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | KRX-0502
Number analyzed (Participants) | 32
g/dL
  Baseline | 10.8 (0.77)
  Week 8 | 11.1 (0.81)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | KRX-0502
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 25/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRX-0502 (N=32)
Rib Fracture (General disorders) | 1
Urinary Tract Infection (General disorders) | 1
General Physical Health Deterioration (General disorders) | 1
Cardiac Failure Chronic (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KRX-0502 (N=32)
Diarrhoea (Gastrointestinal disorders) | 9
Faeces Discoloured (Gastrointestinal disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 3
Abdominal Discomfort (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Weight Decrease (Investigations) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 2
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days